CLINICAL TRIAL: NCT03819517
Title: Improving Cardiovascular Health in Patients With Chronic Obstructive Pulmonary Disease: a Mechanistic Approach
Brief Title: Improving Cardiovascular Health in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HM20014536
Record Dates: First submitted 2018-12-12; First posted 2019-01-28 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Active Comparator): 500 mg of time released micronized trans-Resveratrol
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Placebo will be used in the form of an empty white colored soft vegetarian capsule as resveratrol is presented
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Resveratrol — Over the counter supplementation
  Arms: Resveratrol
Other: Placebo — Empty white colored soft vegetarian capsule
  Arms: Placebo

SUMMARY:
Researchers have found a link between chronic obstructive pulmonary disease (COPD) and heart disease; however, a link is all they have found. Cardiovascular health in COPD is controlled by different mechanisms including vascular health and systemic inflammation. The investigators have collected preliminary data to support that concentrations of Sirtuin 1 (Sirt1), a protein that plays a key role in cardioprotection, may be involved in cardiovascular health in patients with COPD. Resveratrol, an over the counter natural polyphenol found in a variety of food, is a direct activator of Sirt1 and has been used to improve cardiovascular health in different cohorts. The current project is an attempt to expand previous findings and explore the effects of the sub-chronic use of resveratrol in sustaining the improvements in cardiovascular health in COPD.

DETAILED DESCRIPTION:
The present study is designed as a double-blind, randomized, cross-over, placebo-controlled protocol. Patients with COPD will receive either resveratrol (500 mg) or placebo for 12 weeks. A comprehensive evaluation of cardiovascular health will be performed. Results will provide novel insights into the mechanistic role that Sirt1 mediates in COPD related vascular dysfunction and systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a clinical diagnosis of COPD known for at least one year will be allowed to participate
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) stages II to IV
* Breathing test ratio (FEV1/FVC) <0.7
* Amount of exhaled air (FEV1) <80% predicted after bronchodilator
* Total Lung Capacity (TLC)>80%
* Matched healthy volunteers without COPD.

Exclusion Criteria:

* FEV1/FVC>0.7
* Clinical diagnosis of heart disease, hypertension or diabetes
* Use of vasoactive medications (nitrates, Beta blockers)
* Uncontrolled high blood pressure
* Pulmonary hypertension
* Fluid in the lungs
* Sleep apnea
* Thyroid problems
* Anemia
* Raynaud's phenomenon
* Gastrointestinal bleeding
* History of coagulopathies
* History of low platelets
* Gangrene of the digits
* Phenylketonuria
* Pregnant or women attempting to become pregnant
* In lactation
* Individuals who may not be able to read or understand the resveratrol label

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Sirt1 concentrations | Baseline to 12 weeks
  Circulating concentrations of Sirt1 before and 12 weeks after both resveratrol and placebo
Change in vascular health | Baseline to 12 weeks
  Assessment of vascular health through the evaluation of peripheral vascular using the flow-mediated dilation technique before and 12 weeks after both resveratrol and placebo.
Change in Systemic Inflammation | Baseline to 12 weeks
  Systemic inflammation will be evaluated through the assessment of interleukin concentrations using enzyme-linked immunosorbent assay before and 12 weeks after both resveratrol and placebo.

SECONDARY OUTCOMES:
Change in Nitric Oxide metabolism | Baseline to 12 weeks
  Nitric oxide metabolism will be evaluated through Nitric oxide synthase expression using western blot analysis
Change in Inflammatory activation | Baseline to 12 weeks
  The inflammatory cascade of the nuclear factor kappa B will be evaluated through assessment of p65 and p50 expression using western blot analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodriguez Miguelez, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No